CLINICAL TRIAL: NCT06668454
Title: Chemoimmunotherapy Followed by Surgery for Oligometastatic Esophageal and Gastric Cancer: A Phase II Clinical Trial (TORO Protocol)
Brief Title: Chemoimmunotherapy Followed by Surgery for Oligometastatic Esophagogastric Cancer: (TORO Protocol)
Acronym: TORO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTO Project 4717
Record Dates: First submitted 2024-10-25; First posted 2024-10-31 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Esophageal Cancer; Gastric Cancer; Oligometastatic Disease
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surgical Arm (Other): Surgical resection followed by preoperative chemoimmunotherapy for oligometastatic esophagogastric cancer
  Interventions: Procedure: Surgical resection followed by preoperative chemoimmunotherapy for oligometastatic esophagogastric cancer

INTERVENTIONS:
Procedure: Surgical resection followed by preoperative chemoimmunotherapy for oligometastatic esophagogastric cancer — Surgical resection followed by preoperative chemoimmunotherapy for oligometastatic esophagogastric cancer

SUMMARY:
Esophageal cancer and cancers of the gastroesophageal junction (GEJ) are among the most common malignancies worldwide. The outcome for these patients remains very poor. Patients with limited spread of their cancer (oligometastatic disease) have a better prognosis than those with widespread disease. Recent advances in treatment therapies, including use of pre-operative immunotherapy, surgery and/or targeted radiation (SBRT) may help to prolong lifespan in patients with oligometastatic disease. Patients will undergo treatment for their oligometastatic esophageal or gastric cancer with pre-operative chemoimmunotherapy followed by surgery and possibly SBRT to evaluate the value of adding surgery and possibly SBRT to their treatment.

DETAILED DESCRIPTION:
Esophageal cancer and cancers of the gastroesophageal junction (GEJ) are among the most common malignancies worldwide, and the prognosis for patients with metastatic disease remain very poor. However, recent advances in systemic treatment modalities have shown promise for patients with oligometastatic disease, in particular with the incorporation of immunotherapy an targeted agents into systemic treatment regimens. The definition of oligometastatic disease varies across studies and primary sites, but it is generally agreed that patients with oligometastatic disease have a more favorable prognosis than those with widespread metastases. For patients with oligometastatic disease, which is variably defined as the presence of a limited number of metastases, the role of local treatment remains controversial. Chemoimmunotherapy followed by surgery has emerged as a potential treatment option for oligometastatic esophageal and gastric cancer, but further research is needed to evaluate its efficacy and safety and to provide prospective survival and recurrence information.

Several studies have investigated the use of surgery for oligometastatic esophageal cancer after chemo-immunotherapy. A retrospective study of 47 patients with oligometastatic esophageal cancer who underwent immunotherapy and surgery found that the median overall survival was 22 months, and the 2-year overall survival rate was 47.8%. A phase II study of chemoimmunotherapy followed by surgery for patients with oligometastatic esophageal cancer found that the 2-year progression-free survival rate was 60%, and the median overall survival had not been reached at the time of analysis. These studies suggest that surgery after immunotherapy may be associated with better survival outcomes for patients with oligometastatic esophageal cancer, but further research is needed to confirm these findings. SBRT has been evaluated previously in oligometastatic disease in a number of different settings, including in our own institution in studies that included esophageal cancer patients, although in very small numbers. These studies were encouraging but a more thorough evaluation in combination with surgical resection has not been completed.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-proven cT1-4aN0-3M1 adenocarcinoma or squamous cell carcinoma of the esophagus, or EGJ according to the 8th edition of the Union for International Cancer Control (UICC) TNM classification for Esophageal Cancer;
* Oligometastatic disease, which is defined as a maximum of five metastatic lesions, that is treatable by surgical resection or radiation. These five lesions can be present in a maximum of two organs (eg, liver, lung or adrenal gland). Lymph nodes are not counted as an organ. If metastatic retroperitoneal or supraclavicular lymph nodes are present, this lymph node site counts as one metastatic lesion, and together with the possible metastases in organs cannot exceed the number of five lesions.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1;
* Adequate cardiac and respiratory function by standard electrocardiogram and additional diagnostics in case of cardiopulmonary complaints or comorbidity (i.e. lung function test, or echocardiography)
* Adequate blood work parameters for systemic therapy as per treating medical oncologist in terms of ANC, platelet count and hemoglobin.
* Adequate renal function (glomerular filtration rate >50 mL/min or serum creatinine ≤1.5x upper level of normal (ULN)) and adequate liver function (total bilirubin < 2.5x ULN and alanine transaminase (ALT) < 3x ULN);
* A negative serum pregnancy test in women of child-bearing potential during screening period.
* Age >18 and <80 years old

Exclusion Criteria:

* Patients with overt peritoneal or pleural dissemination, as detected on PET-CT or regular CT-scan. In patients in whom a diagnostic laparoscopy is indicated (to assess gastric involvement and the possibility to perform gastric tube reconstruction or to exclude peritoneal disease), tumor-positive cytology peritoneal fluid is also an exclusion criteria. Of note, positive microscopic peritoneal cytology which converts to negative after treatment is not an exclusion criteria (i.e. peritoneal or pleural fluid cytology must be negative at the time of enrollment, with no gross disease identified initially).
* Multiple bone or brain metastases - up to one solitary bone met and/one solitary brain met is allowable as a metastatic site, if curative ablative radiotherapy can be given at the discretion of the treating physicians. Patients with multiple brain metastases or multiple bone metastases will be excluded.
* Any other condition that, in the opinion of the investigator, would make the patient unsuitable for the study; particularly any condition that would make the patient unfit for surgery, radiation, chemotherapy or a combination thereof.
* Active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs) except vitiligo or resolved childhood asthma/atopy. Replacement therapy, such as thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, is not considered a form of systemic treatment and is allowed. Use of non-systemic steroids is permitted.
* Patients with active pregnancy, or lactation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-05-09 (Actual); Primary Completion 2035-05-09 (Estimated); Study Completion 2035-05-09 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 years
  Overall survival outcomes for patients undergoing systemic treatment, primarily with chemoimmunotherapy, followed by surgery in patients with oligometastatic esophageal and GEJ cancer

SECONDARY OUTCOMES:
Surgical safety | Within first 30 days after surgery
  Review of surgical safety, defined by surgical complications
Mortality | Within first 30 days after surgery
  Review of surgical safety, defined by mortality within the first 30 days
Progression free survival | 2 years and 5 years
  Review of distant and loco-regional recurrence
Quality of Life questionnaires | Pre-treatment, post-chemoimmunotherapy/pre-op, post op visit @ 30 days, 6 months, 1 year, 18 months and 2 and 5 years
  Use of FACT E questionnaires at different timepoints to assess patient reported outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Elliot Wakeam, Principal Investigator — Toronto General Hospital-UHN
Locations (1):
- Toronto General Hospital, University Health Network, Toronto, Ontario, Canada